CLINICAL TRIAL: NCT06082882
Title: A Community Based Program to Increase Breast and Cervical Cancer Screening and HPV Vaccination to Reduce the Impact of Breast and Cervical Cancer Among Latinas.
Brief Title: Salud en Mis Manos - Breast and Cervical Cancer Prevention and Early Detection - Expansion 2
Acronym: SEMM2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Cancer Prevention Research Institute of Texas (Other)
Responsible Party: Principal Investigator, Lara Savas, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HSC-SPH-19-0775; PP190061 (Other Grant/Funding Number: Cancer Prevention and Research Institute of Texas)
Record Dates: First submitted 2023-10-09; First posted 2023-10-13 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Breast Cancer; Cervical Cancer
Keywords: Cervical cancer screening; Breast cancer detection; HPV vaccination
MeSH Terms: conditions — Breast Neoplasms; Uterine Cervical Neoplasms | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- In-Person Delivered Breast and Cervical Cancer Behavioral Intervention (Experimental): Community health worker delivered behavioral education and referrals to low-cost services. Delivered in person to participants in community and clinic settings. Participants are followed up by health coach navigators to address barriers and connect to safety-net clinics.
  Interventions: Behavioral: Education; Behavioral: Navigation to clinic
- Telephone Delivered Breast and Cervical Cancer Behavioral Intervention (Experimental): Community health worker delivered behavioral education and referrals to low-cost services. Delivered by telephone to individual participants. Participants are followed up by health coach navigators to address barriers and connect to safety-net clinics.
  Interventions: Behavioral: Education; Behavioral: Navigation to clinic
- Zoom Delivered Breast and Cervical Cancer Behavioral Intervention (Experimental): Community health worker delivered behavioral education and referrals to low-cost services. Delivered by Zoom to individual participants. Participants are followed up by health coach navigators to address barriers and connect to safety-net clinics.
  Interventions: Behavioral: Education; Behavioral: Navigation to clinic

INTERVENTIONS:
Behavioral: Education — Education will be delivered in person in a group education setting or individually by phone. Group education will include a ~1-hour breast and cervical cancer prevention education session delivered with the support of electronic presentations (e.g. PowerPoint presentation ) which will include updated prevention recommendations, such as HPV vaccination recommendations for young adults. For phone education, trained project staff or CHWs will deliver telephone-based education as an alternative to group education sessions for women who missed a scheduled session twice (education materials would be printed and mailed).
Behavioral: Navigation to clinic — Continue telephone based navigation tailored to participants' barriers using the SEMM Cancer Prevention Plan of Action to support, problem solve, assist, and provide reminders to increase utilization of clinic services.

SUMMARY:
The purpose of this study is to increase early detection and prevention of breast and cervical cancer through education and navigation and to increase breast and cervical cancer screening and Human Papillomavirus (HPV) vaccination in underserved Latinas.

DETAILED DESCRIPTION:
This is an evaluation of the implementation of the Salud en Mis Manos program. The investigators evaluate the effect of the program on increasing participant breast and cervical cancer screening and HPV vaccination using a one-group pre-post study design (2022-2024). The investigators also describe the implementation of the program during a longer time period (2020-.2024).

ELIGIBILITY:
Inclusion Criteria:

* Primarily residing in the Gulf Coast & Lower Rio Grande Valley county areas (or other counties in Texas)
* Women 40 years of age and older with no mammogram in the past 2 years
* Women 21-65 years, with no Pap test in the past 3 years
* Women aged 18-26 years, who have not initiated or completed the HPV vaccine series, and through age 45 years if Advisory Committee on Immunization Practices (ACIP) recommends the FDA-approved age expansion for HPV vaccination for older individuals.

Exclusion Criteria:

* Current pregnancy
* Have a current or prior cancer diagnosis

Ages: 18 Years to 74 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8000 (Estimated)
Dates: Start 2020-02-20 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Number of women 40 and older who complete mammogram screening | Between baseline and end of study (about 9 months)
  Among women 40 and older enrolled in the program who have not had a mammogram in the past 2 years at baseline and who self-report mammogram screening completed on follow-up surveys
Number of women 21-65 years who complete Pap test screening | Between baseline and end of study (about 9 months)
  Among women 21-65 years enrolled in the program who have not had a Pap test screening in the past three years at baseline, and who self-report Pap or HPV screening on follow-up surveys.
Number of women 18-26 years who initiate (complete first dose) of the HPV vaccine | Between baseline and end of study (about 9 months)
  Among women 18-26 years that have not had any HPV vaccination at baseline, enrolled in the program and self-report first HPV vaccine completed on follow-up surveys.

SECONDARY OUTCOMES:
Number of women 18-26 years who receive dose 2 of HPV vaccine | between baseline and end of study (about 9 months)
  Among women 18-26 years that have not had their second HPV vaccination dose at baseline, enrolled in the program and self-report completed 2 doses on follow-up surveys.
Number of women 18-26 years who receive dose 3 of HPV vaccine | between baseline and end of study (about 9 months)
  Among women 18-26 years that have not had their third HPV vaccination dose, enrolled in the program and completed baseline and follow-up surveys.

CONTACTS AND LOCATIONS:
Overall Officials: Lara Savas, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No